CLINICAL TRIAL: NCT00207662
Title: ACCENT I - A Randomized, Double-blind, Placebo-controlled Trial of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab, Remicade) in the Long-term Treatment of Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Safety and Efficacy Study of Infliximab (Remicade) in Patients With Moderate to Severe Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004771
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab or placebo

SUMMARY:
This is a study of infliximab (Remicade) in subjects with Crohn's disease

DETAILED DESCRIPTION:
Crohn's disease is a disease characterized by inflammation (the changes that happen when tissues in the body are injured) and ulceration (formation of pus) of the bowel. The purpose of this study is to investigate the safety and therapeutic effect of two different doses of an anti-TNFα (tumor necrosis factor) antibody (a protein) given multiple times compared to a single dose followed by placebo (inactive substance). The name of the antibody is infliximab (Remicade) The goal of the study is to evaluate whether patients respond longer to a single dose of infliximab or to repeated doses of infliximab.

Subjects will receive an infusion of infliximab at week 0 followed by infusions of infliximab or placebo at weeks 2, 6, 14 and every 8 weeks until week 54. Patients who lose response are eligible for additional infliximab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >=18 years of age
* Diagnosis of Crohn's
* Crohn's disease of at least 3 months duration, with colitis, ileitis, or ileocolitis, confirmed by radiography or endoscopy

Exclusion Criteria:

* Local manifestations of Crohn's disease such as strictures, abscesses, or other disease
* Surgery for bowel diversion with placement of a stoma within 3 months prior to beginning the study
* Positive stool culture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2000-07; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Reductions in the signs and symptoms of Crohn's disease

SECONDARY OUTCOMES:
Clinical remission;reduction in the use corticosteroids; mucosal healing

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Rutgeerts P, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Hanauer SB. Comparison of scheduled and episodic treatment strategies of infliximab in Crohn's disease. Gastroenterology. 2004 Feb;126(2):402-13. doi: 10.1053/j.gastro.2003.11.014. PMID 14762776
- [Result] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Derived] Reinisch W, Wang Y, Oddens BJ, Link R. C-reactive protein, an indicator for maintained response or remission to infliximab in patients with Crohn's disease: a post-hoc analysis from ACCENT I. Aliment Pharmacol Ther. 2012 Mar;35(5):568-76. doi: 10.1111/j.1365-2036.2011.04987.x. Epub 2012 Jan 18. PMID 22251435